CLINICAL TRIAL: NCT06713850
Title: Real-World Clinical Evaluation of the Shockwave Intravascular Lithotripsy (IVL) Catheter System for Treating Severe Calcified Lesions in Femoropopliteal Arteries
Brief Title: Angioplasty With Shockwave IVL Catheter System in Femoropopliteal Lesions
Acronym: SHIELD
Status: Recruiting | Type: Observational
Sponsor: Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Huashan Hospital (Other); Xuanwu Hospital, Beijing (Other); The General Hospital of Southern Theater Command (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); RenJi Hospital (Other); Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zibo Feng, Professor, Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: the SHIELD study
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Artery Disease (PAD); Chronic Limb Threatening Ischemia
Keywords: Peripheral Artery Disease; Chronic Limb Threatening Ischemia; Severe calcification
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Shockwave balloons — To evaluate the effectiveness and safety of the Shockwave intraperipheral shockwave catheter system in peripheral arterial angioplasty.

SUMMARY:
There is a lack of prospective observational studies of shockwave balloons in the treatment of moderate-to-severe calcification of the femoral popliteal artery at the international level. Therefore, in this study, we wish to set up a real-world study of shockwave balloon in the treatment of moderate-to-severe calcification to investigate the real-world efficacy of shockwave balloon in the treatment of moderate-to-severe calcified lesions.

DETAILED DESCRIPTION:
Vascular calcification is prevalent in patients with peripheral artery disease (PAD), especially those with comorbid diabetes or chronic kidney disease. Severe calcification portends a poor prognosis and is independently associated with an increased risk of cardiovascular mortality and morbidity. Calcification may also compromise the efficacy of endoluminal therapy, leading to suboptimal vasodilatation and an increased risk of vascular complications, including restenosis, as well as entrapment, perforation, and distal embolization. The current grading of vascular calcification is based on the PACSS score, which can be categorized as mild, moderate, or severe depending on the degree of calcification and the extent of the lesion. Neither high-pressure balloon angioplasty nor plaque resection (atherectomy) significantly improves severely calcified lesions. The efficacy of these treatment modalities has also not been validated in multicenter real-world studies. Shockwave balloons have been widely used in the clinical endoluminal treatment of severely calcified lesions due to their ability to significantly disrupt calcified structures while reducing damage to the vascular intima, thereby reducing postoperative complications. The current published study Disrupt PAD III Trial (NCT02923193) of shockwave balloon treatment of calcified lesions demonstrated a lower residual stenosis rate with shockwave balloon versus balloon dilatation alone in a randomized controlled trial (RCT) (66.4% vs. 51.9%; p = 0.02), limiting the number of patients who could be treated with shockwave balloon. p = 0.02), a lower incidence of flow-limiting entrapment (1.4% vs. 6.8%; p = 0.03), and a lower rate of posterior dilation and remedial stenting (5.2% vs. 17.0%; p = 0.001); (4.6% vs. 18.3%; p < 0.001). Shockwave balloons have been approved by the Chinese Food and Drug Administration for endoluminal treatment of severe calcification of the femoropopliteal artery, and are currently used only in larger vascular surgery centers because of their short time on the market. On this basis, we asked whether we could set up a real-world study of shockwave balloons for the treatment of moderate-to-severe calcification to investigate the real-world efficacy of shockwave balloons in the treatment of moderate-to-severe calcified lesions.

ELIGIBILITY:
Inclusion Criteria:

-

1) Age ≥ 18 years (2) Rutherford Classification 2-5 3) Stenosis (>70% stenosis confirmed by digital subtraction angiography (DSA) imaging) or occlusion of the femoropopliteal artery, with one healthy patent outflow tract distal to the knee in continuity with a patent outflow tract below the ankle.

(4) Patients who understand the purpose of the study, participate in the experiment voluntarily, sign the informed consent form and are willing to be followed up.

5) The guidewire needs to pass through the lesion; 6) Life expectancy >24 months 7) Moderately severe calcified lesions confirmed by imaging data: 8) For patients who receive intervention in both lower extremities may be enrolled in order of time of intracavitary treatment 9) For combined aortoiliac artery lesions that have undergone endoluminal revascularization to achieve flow recanalization without more than 50% residual stenosis.

Exclusion Criteria:

1. Patients with stroke, cerebral hemorrhage, gastrointestinal hemorrhage, or cardiac infarction within 3 months prior to enrollment (2) Patients with known allergy to heparin, aspirin, other antiplatelet drugs, contrast agents, etc.

3) Patients who have been enrolled in medications that interfere with this clinical trial within the last 3 months or who have been treated intraoperatively with other special vascular bed preparation devices, such as plaque volume reduction devices, special balloons, and so on; 4) Pregnant and lactating women 5) Patients who are unable or unwilling to participate in this trial. 6) patients with Berger's disease 7) patients who have received arterial bypass diversion on the treated side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PAD.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Procedural Success Rate | procedural
  Residual stenosis <50% with no flow-limiting entrapment after study device therapy (before subsequent endovascular device therapy).

SECONDARY OUTCOMES:
Primary Patency Rate | 30 days
  Primary patency of target lesions at 30 days postoperatively
Freedom from clinically-driven target lesion revascularization(CD-TLR) | 1 month, 3 months, 6 months, 12 months
  Clinically driven target lesion revascularization is defined as target lesion revascularization performed due to target lesion diameter stenosis ≥50% and either evidence of clinical or functional ischemia (e.g., recurrent/progressive life-limiting intermittent claudication, claudication unresponsive to medical therapy, CLI) or recurrence of the clinical syndrome for which the initial procedure was performed.
Clinical improvement | 1 month, 3 months, 6 months, 12 months
  Improvements in Rutherford grading
Vascular quality of life questionnaire(VascuQol) | 1 month, 3 months, 6 months, 12 months
  The VascuQol was designed as a questionnaire containing five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items) to evaluate Health related quality of life (HRQL). Every item has seven response options, with scores ranging from 1 to 7. A total score is the sum of all 25 item scores divided by 25.And both the total score as well as the domain scores range from 1 (worst HRQL) to 7 (best HRQL).The lower the value, the poorer the quality of life.
Remedial stenting rate | procedural
  Remedial stenting rate
Remedial stenting rate | 1 month, 3 months, 6 months, 12 months
  Manipulation-related acute thrombosis, arterial embolism, major amputation, and all-cause mortality
Instrument success | procedural
  Successful delivery and deployment of a single-use peripheral intravascular shockwave catheter to the intended target lesion site and successful withdrawal of the delivery system
Incidence of Major Adverse Events at 30 days postoperatively | 30 days
  a Emergency surgical hemodialysis of the target limb; b.Unplanned target limb amputation (above the ankle); c.Symptomatic thrombosis or distal embolization requiring treatment in the area of the target lesion or in the target limb as confirmed by imaging; d.Perforation or flow-limiting entrapment of the target lesion requiring treatment; cardiac death.
Major adverse events | 1 month, 3 months, 6 months, 12 months
  Death, unplanned major amputation of the target limb, and CD-TLR were defined as a major adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
This is a multi-center real-world study and the data will be shared among several of the participating centers. For non-participants who need to use the data, consent from all participating units will be required before use.